CLINICAL TRIAL: NCT04718753
Title: Positive Spiral of Mindfulness in Mindful Breathing: A Pilot Randomized Controlled Trial Using Ecological Momentary Assessment and Actigraphy
Brief Title: Mindful Breathing Using EMA and and Actigraphy: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSY013
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Mindfulness
Keywords: Mindfulness; Mindful breathing; Positive spiral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Breathing Group (Experimental): Mindful breathing intervention which has been used in mindfulness-based interventions
  Interventions: Behavioral: Mindful breathing intervention
- Waitlist Control Group (No Intervention): Participants in the waitlist control group will receive the intervention after the immediate post-treatment assessment

INTERVENTIONS:
Behavioral: Mindful breathing intervention — Mindful breathing intervention audio, which is used in mindfulness-based interventions, will be sent to the participants once per day.
  Arms: Mindful Breathing Group

SUMMARY:
This study will examine the effect of mindful breathing and the mechanism of positive spirals of mindfulness using ecological momentary assessment (EMA) and actigraphy. Previous studies have shown a positive spiral between state mindfulness and positive affect (Du, An, Ding, Zhang, & Xu, 2018). The mindful coping model (Garland, Gaylord, & Fredrickson, 2011) suggested that the state of mindfulness can lead to reappraisal and reframing of their stressful circumstances which further lead to positive emotion and reduced stress. These positive effects will affect the next cycle and hence form a positive spiral. Since mindful breathing was an effective practice for immediate decentering (Feldman, Greeson, & Senville, 2010), it will be used as the manipulation of state mindfulness. Besides, there is very limited research on the associations between these constructs using EMA and actigraphy. Therefore, this study will explore this association by manipulating the state of mindfulness with mindful breathing using EMA.

DETAILED DESCRIPTION:
This proposed study will be a randomized control trial which studies the mechanism of positive spirals of mindfulness in mindful breathing. Potential participants will be recruited from the community through posters, social media sites and/or emails. About 30 eligible participants will be recruited after an online screening (with phone support). Prior to all study procedures, the research purpose and data collection procedure will be given to the participants and an online informed consent will be obtained from them.

In this study, participants will be randomly assigned to either the mindful breathing group (intervention group) or the waitlist group (control group) in a ratio of 1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. No deception is necessary.

All participants will be requested to wear an actigraphy device (ActiGraph GT9X link) connected to a heart rate sensor (Polar H10) for 8 consecutive days, for recording their physiological data including HRV and activity level. Ecological momentary assessment (EMA) will also be used. A smartphone application will be developed and installed in the participants' smartphones. The app will prompt the participants, 4 times each day (9 a.m., 1 p.m., 5 p.m. and 9 p.m.), to fill in a self-report questionnaire concerning mood. Besides that, participants have to complete an assessment at baseline and immediate post-intervention assessments.

Participants in treatment group will receive mindful breathing instructions daily (at 9 a.m. after completing the EMA questionnaires). They will be asked to perform a 10-minute mindful breathing exercise based on an audio. After that, they will submit a simple record indicating the time they have completed the exercise. Meanwhile, participants in the waitlist condition will not receive the recording during the study. However, the same set of mindful breathing instruction audio will be sent to the waitlist group after the study.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged ≥ 18 years and ≤ 65 years;
2. Cantonese language fluency; and
3. A willingness to provide informed consent and comply with the study protocol.

Exclusion Criteria:

1. Major medical or neurocognitive disorders that make participation infeasible;
2. Having psychiatric disorders based on General Health Questionnaire (GHQ-28) score > 11 or having suicidal ideation based on a positive answer to question 27 and 28 (referral information to professional services will be provided to those who endorsed items on suicidal ideation);
3. Cardiovascular diseases that affect the measure of heart rate variability (HRV); and
4. Using medication or psychotherapy for any psychological disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Ecological momentary assessment (EMA) - Mindful Attention Awareness Scale (MAAS) | Baseline (1day), intervention/ waitlist period (four times per day over 7days) and immediately post-intervention (7days)
  An in-house smartphone application will be developed and installed in the participant's smartphones for recording the participants' mindfulness at baseline once and 4 times a day over 7 consecutive days. MAAS is a 15-item scale widely used to assess the level of mindfulness, which scores each of the 15 statements as "1" (almost always) to "6" (almost never). The computed score is calculated by averaging the 15 scores. State MAAS is a 5-item scale developed from MAAS, which scores each of the 5 statements as "0" (almost always) to "6" (almost never). The MAAS will be used in baseline and immediately post-intervention while the state MAAS will be used in baseline and intervention/ waitlist period via EMA.
Change in EMA - Positive and Negative Affect Scale (PANAS) | Baseline (1day), intervention/ waitlist period (four times per day over 7days) and immediately post-intervention (7days)
  An in-house smartphone application will be developed and installed in the participant's smartphones for recording the participants' positive and negative affect at baseline once and 4 times a day over 7 consecutive days. PANAS is a 20-item five-point Likert scale widely used to assess positive and negative mood or emotion. This scale consists of 10 items measuring positive affect and 10 items measuring negative affect.

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scales (DASS-21) | Baseline and immediately post-intervention (7days)
  DASS-21 is a 21-item scale, comprises three sub-scales which measures the negative emotional states of depression, anxiety, and stress, over the past week.
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline and immediately post-intervention (7days)
  The PSQI is a widely used 24-item scale used to access the sleep quality and disturbances over a 1-month interval. The 19 self-rated questions will be used and modified for a 1-week time interval in this study.
Self-developed Survey | Baseline
  The self-developed survey will collect information including demographic information (e.g., age, gender, level of education, working industry, relationship status, and location of residence).
Record of mindful breathing | Intervention period (once a day over 7days)
  The record will collect the time when the participant practice mindful breathing.
Change in Actigraphy (Actigraph GT9X Link; USA Philips Respironics Inc.) - sleep-onset latency (SOL) | Baseline and intervention/ waitlist period (7 days)
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 7 consecutive days, SOL is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actigraph GT9X Link; USA Philips Respironics Inc.) - wake after sleep onset (WASO) | Baseline and intervention/ waitlist period (7 days)
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 7 consecutive days, WASO is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actigraph GT9X Link; USA Philips Respironics Inc.) - total wake time (TWT) | Baseline and intervention/ waitlist period (7 days)
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 7 consecutive days, TWT is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actigraph GT9X Link; USA Philips Respironics Inc.) - total sleep time (TST) | Baseline and intervention/ waitlist period (7 days)
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 7 consecutive days, TST is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actigraph GT9X Link; USA Philips Respironics Inc.) - sleep efficiency (SE) | Baseline and intervention/ waitlist period (7 days)
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 7 consecutive days, SE is one of the sleep parameters which will be measured by Actigraphy.
Change in Polar H10 heart rate sensor (Polar Electro, Inc.) - heart rate variability (HRV) | Baseline and intervention/ waitlist period (7 days)
  Participants will be instructed to wear a wrist-worn actigraphy device and a heart rate sensor strapped around their chest to record their physiological patterns for 7 consecutive days. Heart rate variability (HRV) will be measured by the sensor to indicate stress level.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong